CLINICAL TRIAL: NCT04690348
Title: Intracavitary Carrier-embedded Cs131 Brachytherapy for Recurrent Brain Metastases: a Randomized Phase II Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: GT Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-542
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Brain Metastases
Keywords: Cs-131 Brachytherapy; Brain Metastasis; 20-542
MeSH Terms: conditions — Brain Neoplasms | interventions — Craniotomy

STUDY DESIGN:
Intervention Model Description: Prospective randomized phase II multicenter trial.
Who Masked: Participant
Masking Description: Patient will be blinded to their treatment until postoperatively.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Resection without brachytherapy (Active Comparator): Patients will undergo craniotomy.
  Interventions: Procedure: Craniotomy
- Resection plus brachytherapy (Experimental): Patients will undergo craniotomy and patients in the treatment arm will undergo implantation of Cesium 131 brachytherapy in coordination with the radiation oncologist.
  Interventions: Procedure: Craniotomy; Radiation: Cesium-131 brachytherapy

INTERVENTIONS:
Procedure: Craniotomy — Craniotomy
Radiation: Cesium-131 brachytherapy — Intracavitary Cesium-131 brachytherapy
  Arms: Resection plus brachytherapy

SUMMARY:
The purpose of this study is to see if Cs-131 brachytherapy is effective in people with recurrent brain cancer who are scheduled to have brain surgery for removal of their tumor(s). The researchers would like to see whether Cs-131 prevents brain tumors from growing back after surgery.The researchers will compare Cs-131 brachytherapy (which occurs during brain surgery) with the usual approach of brain surgery without brachytherapy. The researchers will compare both the effectiveness and safety of the two approaches.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age who are capable of giving consent
* Undergoing elective craniotomy for resection of a previously-irradiated brain metastasis with suspicion for viable disease at the time of consent, and anticipated achievement of gross-total or near-total (>/=95%) resection
* Karnofsky Performance Status score (KPS) of ≥70
* Ability to undergo brain MRI with gadolinium

Exclusion Criteria:

* Unable to tolerate MRI or CT imaging
* Pregnancy (patients must have a negative pregnancy test within 30 days of the operation)
* Women must agree to not breastfeed for at least 12 weeks after the procedure (lactating and discarding in that interval allowable)
* Diagnosis of leptomeningeal carcinomatosis or >5 additional active or untreated CNS lesions for a total of >6 active lesions
* Prior irradiation (EQD2) in excess of 100 Gy to site of implant, using an α/β of 2
* Apposition of tumor margin to brainstem or optic apparatus
* Previous infection within the operative field, current active systemic infection requiring systemic therapy, or immunodeficiency
* Urgent surgery required prior to availability of brachytherapy

Intraoperative Exclusion Criterion:

* Patients will be excluded if intraoperative pathology is not consistent with >/=5% viable metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2020-12-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
freedom from local progression | 9 months following surgery
  With a contrast enhanced brain MRI scan. Treatment response will be determined based on the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria.

SECONDARY OUTCOMES:
wound complications | 3 months
  Physical examination including wound examination will be performed, and wound complications (including dehiscence, superficial/deep infection, CSF leak) will be recorded by the evaluating clinicians.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Moss, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Baptist Health South Florida, Miami, Florida
  - Memorial Sloan Kettering at Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm